CLINICAL TRIAL: NCT06528275
Title: Food Insecurity During Pregnancy in French Guiana - Focus on Infant Feeding
Brief Title: Infant Feeding in French Guiana
Acronym: ANJE Nutri
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: ANJE Nutri
Record Dates: First submitted 2024-07-23; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Food Insecurity; Pregnancy Related
Keywords: Infant feeding; Breastfeeding; Food insecurity; Pregnancy; French Guiana
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - control: Pregant women included in Nutri Pou Ti Moun 1 project who did not benefit from the health promotion intervention
- Group 2 - intervention: Pregant women included in Nutri Pou Ti Moun 1 project who benefited from the health promotion intervention
  Interventions: Other: Health promotion intervention

INTERVENTIONS:
Other: Health promotion intervention — Health promotion intervention with activites linked to nutrition, and distribution of baskets of fresh fruits and vegetables
  Groups: Group 2 - intervention

SUMMARY:
This is a comparative, observal study among the population of pregant women who participated to the study "Nutri Pou Ti Moun" on food insecurity during pregnancy in French Guiana

DETAILED DESCRIPTION:
The international literature has already demonstrated the benefits of breastfeeding (BF) in the short, medium and long term for the health of children and mothers alike. For children, breastfeeding helps to reduce mortality from infections, prevents hospitalisations, particularly for gastroenteritis and respiratory illnesses, and prevents diabetes and childhood obesity. Breastfeeding also plays an important role in children's cognitive development, with an impact on IQ and academic success. For mothers, not breastfeeding is associated with an increased risk of breast and ovarian cancer, type II diabetes, obesity and cardiovascular disorders. Similarly, the WHO recommends optimal feeding practices for infants up to 2 years of age, i.e. early initiation of breastfeeding to allow the child to receive colostrum, exclusive BF for 4 to 6 months, and the timely introduction of liquid, semi-solid or solid foods, the continuation of BF for up to 2 years and beyond, the consumption of age-appropriate infant formula (IF) as an alternative to breastfeeding, and a minimum acceptable intake of complementary food to breast or infant milk.

On a national scale, the 'first 1000 days' initiative (from the 4th month of pregnancy to the child's 2nd birthday) that emerged at the symposium on 23 September 2021 organised by Santé Publique France and the French Ministry of Solidarity and Health includes the objective of promoting good BF practices. Similarly, the 2019-2023 national nutrition and health plan (PNNS4) aims to increase the percentage of children breastfed at birth by at least 15% and to extend the median duration of total breastfeeding by 2 weeks. In French Guyana, the 2023-2028 regional health plan points out that perinatal indicators in the French overseas territories are worse than in mainland France, and that improving mother and child health must involve improving the environment in which children live during their first 1,000 days.

In 2005, an initial retrospective study of breastfeeding practices was carried out in western part of French Guiana and showed a rate of exclusive breastfeeding at 4 months of age of 3% and a rate of continued breastfeeding of 16.7% up to 1 year and 6.5% up to 2 years. Between 2010 and 2012, a prospective survey of the whole of French Guiana found an exclusive BF rate of 27% at 1 month, 9% at 3 months and 5% at 6 months. In the Epifane survey conducted in France between 2010 and 2012, the rate of exclusive breastfeeding at 1 month and 3 months was close to that in French Guiana (28% and 10% respectively), with an average duration of exclusive or predominant breastfeeding of 3 weeks.

The rate of continued breastfeeding for up to 1 year was estimated at 16% in the Guiana study, compared with 9% in France. The rate of mixed breastfeeding concerned 30% of women breastfeeding from the maternity hospital in French Guiana, compared with 20% in France. The main reasons for introducing bottles of infant formula (IF) in both French Guiana and France were the impression of a lack of milk (the child's feeling of dissatisfaction) and the return to work. On the other hand, almost 1 in 2 women in French Guiana stated that no healthcare professional had shown any interest in their breastfeeding at 1 month post-partum.

Since January 2023, the Nutri Pou Ti'moun study ('Nutri 1 project' ID-RCB 2022-A01772-41), carried out in 3 maternity units in French Guiana and involving 800 women who have given birth - the 'Nutri 1 women's group' - aims to take stock of women's food insecurity during pregnancy and to describe the medical consequences observed on the course and outcome of pregnancy and on infant health in the immediate post-partum period. In the course of this project, the links between vitamin and mineral deficiencies, heavy metal impregnation and maternal dietary diversification are being studied. In the Guianese context of multidimensional precariousness, the Guianese perinat network, in partnership with local and institutional players, aimed to set up a health and nutrition pathway from the 4th month of pregnancy in October 2023, comprising weekly workshops co-hosted by a health mediator (on diet, well-being, adapted physical activities and the promotion of breastfeeding) and the distribution of baskets of fresh, local fruit and vegetables.

This health promotion intervention is offered to pregnant women attending the maternal and child health protection centre (PMI) in the Communauté d'agglomération du centre littoral (CACL) - the 'Nutri 2 women's group'. This intervention gave rise to an ancillary research project to the Nutri Pou Ti'moun research project, the Nutri pou ti'moun 2 project (Nutri 2 project; ID-RCB 2023-A00167-38) aimed at assessing the impact of this action on women's diet (diversity and food insecurity) by comparing the data from the Nutri 1 women's group with that from the Nutri 2 women's group. These projects only cover the period from pregnancy to the immediate post-partum period. By 31 December 2023, 786 women had been included in the Nutri 1 project and 57 women in the ancillary Nutri 2 project.

The relevance and interest of conducting research in French Guiana on breastfeeding practices and, more broadly, on infant feeding are justified:

* On the one hand, by the absence of recent published data on infant feeding practices in French Guiana. The second national Epifane survey, to be carried out in 2021 and focusing on infant nutrition during the first year of life, is a study being conducted in parallel with the national perinatal survey in France. An extension of this survey was carried out in the French overseas departments and territories, but French Guiana was not included.
* On the other hand, the Nutri Pou Ti Moun project represents an opportunity to collect data on infant feeding from a representative sample of women giving birth in French Guiana, in the three public maternity hospitals (Nutri 1 group of women). Medical, biomedical and socio-demographic data, as well as data relating to food safety and nutrition during pregnancy already collected during the Nutri Pou Ti moun project, will be analysed with regard to infant feeding practices and child development data (staturo-weight, cranial perimeter, psychomotor development). The impact of a prenatal intervention on nutrition could also be assessed by comparing infant feeding data for children in the Nutri 1 group and those in the Nutri 2 group.

In a socio-economic and health context that is different from that in mainland France, food insecurity in French Guiana during pregnancy, as assessed in the Nutri Pou Ti moun project, is likely to have consequences for young children that it would be relevant to measure and compare with national and international data. In the short term, the impact of this food insecurity would influence the use and duration of breastfeeding, the occurrence of anaemia in young children and dietary practices; and in the medium term, the child's staturo-weight development and cognitive development.

ELIGIBILITY:
Inclusion Criteria:

* Intervention group : women included in Nutri Pou Ti Moun project and who benefited from health promotion intervention
* Control group : women included in Nutri Pou Ti Moun project and who did not benefit from health promotion intervention

Exclusion Criteria:

* Women refusing to participate to the study
* Women who moved out of French Guiana
* Women lost for follow up or who could not be contacted for the participation to the study
* Minor women who could not obtain authorisation from legal representatives

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women living in French Guiana who participated to the Nutri Pou Ti Moun project and who benefited or not from a health promotion intervention on nutrition
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of exclusive breastfeeding at 3 months of age in French Guiana | At inclusion
  To estimate the prevalence of exlusive breastfeeding at 3 months of age in French Guiana in the group control and the group intervention

SECONDARY OUTCOMES:
Description of exclusive breastfeeding practices | At inclusion
  To describe exclusive breasfeeding practices by questionnaire
Description of artificial breastfeeding practices | At inclusion
  To describe artificial breastfeeding practices by questionnaire
Description of dietary diversity in infants | At inclusion
  To describe dietary diversity in infants by questionnaire
Description of the minimal dietary diversity | 12 months
  To describe the minimal dietary diversity for children 6-23 months (MDD-IYCF) at 12 months of age by questionnaire
Description of the minimal dietary diversity of mothers | 12 months
  To describe the minimal dietary diversity of mothers (MDD-W) at 12 months of age of the baby by questionnaire
Description of staturo-ponderal and psychomotor development indicators | 12 months
  Prevalence of staturo-ponderal and psychomotor development indicators among infants during their 1st year of age
Breastfeeding rate, exclusive and artificial breastfeeding duration, dietary diversity between groups | 12 months
  Comparison of breastfeeding rate, exclusive and artificial breastfeeding duration, dietary diversity and age at diversity between the 2 groups
Description of breastfeeding practices from mothers point of view | At inclusion
  To describe views on breastfeeding practices in intervention group by semi-structured interview
Description of breastfeeding practices from professionals point of view | At inclusion
  To describe views on breastfeeding practices in professionals by semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Celia BASURKO, MD, Principal Investigator — Centre Hospitalier de Cayenne
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Sankar MJ, Sinha B, Chowdhury R, Bhandari N, Taneja S, Martines J, Bahl R. Optimal breastfeeding practices and infant and child mortality: a systematic review and meta-analysis. Acta Paediatr. 2015 Dec;104(467):3-13. doi: 10.1111/apa.13147. PMID 26249674
- [Background] Horta BL, Loret de Mola C, Victora CG. Long-term consequences of breastfeeding on cholesterol, obesity, systolic blood pressure and type 2 diabetes: a systematic review and meta-analysis. Acta Paediatr. 2015 Dec;104(467):30-7. doi: 10.1111/apa.13133. PMID 26192560
- [Background] Binns C, Lee M, Low WY. The Long-Term Public Health Benefits of Breastfeeding. Asia Pac J Public Health. 2016 Jan;28(1):7-14. doi: 10.1177/1010539515624964. PMID 26792873
- [Background] Chowdhury R, Sinha B, Sankar MJ, Taneja S, Bhandari N, Rollins N, Bahl R, Martines J. Breastfeeding and maternal health outcomes: a systematic review and meta-analysis. Acta Paediatr. 2015 Dec;104(467):96-113. doi: 10.1111/apa.13102. PMID 26172878
- [Background] Basurko C, Dupart O, Savy M, Obert-Marby C, Mvogo A, Gonzalez A, Trepont A, Cann L, Boceno C, Osei L, Creton PM, Dufit V, Thelusme L, Adenis A, Van-Melle A, Huber F, Nacher M. Hunger in French Guiana's Vulnerable Urban Neighborhoods: A Neglected Consequence of COVID-19. Food Nutr Bull. 2023 Mar;44(1):3-11. doi: 10.1177/03795721231156641. Epub 2023 Feb 23. PMID 36824041
- [Background] Nacher M, Basurko C, Muhigirwa GB, Lambert V, Osei L, Njuieyon F, Louis A, Dotou D, Thomas N, Bernard S, Leneuve M, Elenga N, Hcini N. Infant mortality in French Guiana between 2001 and 2017 : Trends and comparisons with mainland France. Rev Epidemiol Sante Publique. 2023 Dec;71(6):102175. doi: 10.1016/j.respe.2023.102175. Epub 2023 Oct 31. PMID 37918040
- See also: Short-term effects of breastfeeding: a systematic review on the benefits of breastfeeding on diarrhoea and pneumonia mortality — https://iris.who.int/handle/10665/95585
- See also: Indicators for assessing infant and young child feeding practices — https://iris.who.int/bitstream/handle/10665/43895/9789241596664_eng.pdf?sequence=1
- See also: Conference on the "1000 first days" - Santé Publique France - 23 September 2021 — https://www.santepubliquefrance.fr/a-propos/evenements/colloque-les-1000-premiers-jours-23-septembre-2021
- See also: French national health and nutrition program — https://sante.gouv.fr/IMG/pdf/pnns4_2019-2023.pdf
- See also: French Guiana Regional Health Program 2018-2028 — https://www.guyane.ars.sante.fr/revision-du-projet-regional-de-sante-prs-guyane-2018-2028
- See also: Duration of breastfeeding period in France - Epifane survey 2012-2013 — https://beh.santepubliquefrance.fr/beh/2014/27/2014_27_2.html
- See also: French Guiana Regional program on access to prevention and care — https://www.guyane.ars.sante.fr/media/116268/download?inline